CLINICAL TRIAL: NCT03133130
Title: A Randomized, Single Blind, Single Dose, Placebo-controlled, Dose-escalation Phase I Study to Investigate the Pharmacokinetics, Safety, and Tolerability of Intradermal Dosage Form of BMT101 in Healthy Male Volunteers
Brief Title: Study to Investigate the Pharmacokinetics, Safety, and Tolerability of BMT101 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hugel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HG-BMT-PI-01
Record Dates: First submitted 2017-03-28; First posted 2017-04-28 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2017-04

CONDITIONS: Hypertrophic Scar
Keywords: Scar; Scar prevention; siRNA
MeSH Terms: conditions — Cicatrix, Hypertrophic; Cicatrix

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMT101 (Experimental): cp-lasiRNA
  Interventions: Drug: BMT101
- Placebo (Placebo Comparator): Normal Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMT101 — BMT101 is administered to 6 subjects in each of 4 groups.
  Arms: BMT101
Drug: Placebo — Placebo is administered to 2 subjects in each of 4 groups.
  Arms: Placebo

SUMMARY:
Phase I Study to Investigate the Pharmacokinetics, Safety, and Tolerability of BMT101 in Healthy Male Volunteers

DETAILED DESCRIPTION:
A Randomized, Single Blind, Single Dose, Placebo-controlled, Dose-escalation Phase I Study to Investigate the Pharmacokinetics, Safety, and Tolerability of Intradermal Dosage Form of BMT101 in Healthy Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 19 ~ 39 years of age
2. Body Mass Index (BMI) between 19 to 25kg/㎡ (19kg/㎡ ≤ BMI < 25kg/㎡) and weight at least 50kg on the day of screening
3. Medically healthy with no clinically significant findings on vital signs during the screening period
4. Medically healthy with no clinically significant findings on physical examinations during the screening period

Exclusion Criteria:

1. Subjects with clinically significant medical or surgical history described below Clinically significant observations considered as unsuitable based on medical judgement by investigators

   * Skin disorder (psoriasis or contact dermatitis) which may affect absorption of the investigational product, or scar, skin abnormality, history of surgery (excluding simple appendectomy or herniorrhaphy) which can interrupt intradermal injections
2. History of clinically significant allergy, cardiovascular, peripheral vascular, skin, mucocutaneous, ocular, respiratory, musculoskeletal or any other conditions which can be problems for pharmacokinetic evaluation
3. Donated blood or blood components or had been transfused plasma within 60 days prior to the day of screening
4. Tobacco use within 30 days prior to the day of screening

Ages: 19 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The clinical trial is comparative phase I study of the safety, tolerability, and pharmacokinetic characteristics of Investigational products, not to evaluate the efficacy of treatment. Therefore, other treatments or types are not considered and because this clinical trial has experimental aspects that are not verified, this clinical trial is conducted for healthy male volunteers.
Enrollment: 32 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

PRIMARY OUTCOMES:
Safety Evaluation: Severity and frequency of reported adverse events, clinically-relevant changes in physical exams or laboratory testing assessed by medical personnel | 14 days
  Assess severity and frequency of reported adverse events, clinically-relevant changes in physical exams or laboratory testing assessed by medical personnel

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of BMT101 by intradermal injection following single dose: Cmax | 4 days
  Determine peak whole blood concentration (Cmax)
Pharmacokinetics (PK) of BMT101 by intradermal injection following single dose: AUC | 4 days
  Determine area under the whole blood concentration versus time curve (AUC)
Pharmacokinetics (PK) of BMT101 by intradermal injection following single dose: T½ | 4 days
  Determine drug half-life in whole blood (T½)

CONTACTS AND LOCATIONS:
Locations (1):
- Hugel, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No